CLINICAL TRIAL: NCT02618408
Title: Assessment of the Efficacy and Safety of Molindone Hydrochloride Extended-Release for the Treatment of Impulsive Aggression in Pediatric Patients With Attention Deficit/Hyperactivity Disorder in Conjunction With Standard ADHD Treatment
Brief Title: Treatment of Impulsive Aggression in Subjects With ADHD in Conjunction With Standard ADHD Treatment (CHIME 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 810P301
Record Dates: First submitted 2015-11-20; First posted 2015-12-01 (Estimated); Results first posted 2022-11-01 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2020-11

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose SPN-810 (18 mg) (Experimental): Oral
  Interventions: Drug: SPN-810 (18 mg)
- High dose SPN-810 (36 mg) (Experimental): Oral
  Interventions: Drug: SPN-810 (36 mg)
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPN-810 (18 mg) — Subjects were randomized to receive SPN-810 low dose (18 mg) twice each day (BID) with or without food, in the morning and in the evening, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if after noon, the evening dose.
  Arms: Low dose SPN-810 (18 mg)
Drug: SPN-810 (36 mg) — Subjects were randomized to receive SPN-810 high dose (36 mg) twice each day (BID) with or without food, in the morning and in the evening, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if after noon, the evening dose.
  Arms: High dose SPN-810 (36 mg)
Drug: Placebo — Subjects were randomized to receive Placebo twice each day (BID) with or without food, in the morning and in the evening, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if after noon, the evening dose.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy, safety, and tolerability of SPN-810 in the treatment of Impulsive Aggression (IA) in subjects with Attention-Deficit/Hyperactivity Disorder (ADHD) in conjunction with standard ADHD treatment. Approximately 426 subjects aged 6 to 12 years with ADHD and comorbid impulsive aggression will be recruited in this study. The frequency of impulsive aggression behaviors will be assessed as a primary outcome. Additionally, the severity and improvement in impulsive aggression and quality of life measures for the subject and caregiver will be assessed using validated scales.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, 3-arm, parallel-group study, to assess the efficacy, safety, and tolerability of SPN-810 in the treatment of IA in subjects 6 to 12 years old with ADHD, in conjunction with standard ADHD treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects, age 6 to 12 years at the time of screening.
2. Diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Disorders- 5 (DSM-5 confirmed by the Schedule for Affective Disorders and Schizophrenia for School-aged Children - Present and Lifetime Version 2013 (K-SADS-PL 2013).
3. Retrospective Modified Overt Aggression Scale (R-MOAS) score of ≥24 at screening.
4. CGI-S score of at least moderately ill at both Screening and Randomization.
5. Vitiello Aggression Scale score from -2 to -5 at screening.
6. Free of antipsychotic medication for at least two weeks prior to Visit 2.
7. Monotherapy treatment with FDA-approved optimized ADHD medication (psychostimulant or non-stimulant) at an FDA-approved dose for at least one month prior to screening, and willing to maintain that dose throughout the Baseline and Treatment period.
8. α 2- adrenergic agonists (e.g., clonidine and guanfacine) used for any other reason except for monotherapy treatment for ADHD (e.g., aggression or insomnia) must be discontinued at least two weeks prior to Visit 2.
9. Medically healthy and with clinically normal laboratory profiles, vital signs, and electrocardiograms (ECGs).
10. Weight of at least 20 kg.
11. Able and willing to swallow tablets whole and not chewed, cut, or crushed.
12. Written Informed Consent obtained from the subject's parent or legal representative and written Informed Assent obtained from the subject if appropriate.
13. Measurement of compliance ≥ 80% for completion of IA Diary during Baseline Period.

Exclusion Criteria:

1. Body Mass Index (BMI) in 99th percentile or above.
2. Current or lifetime diagnosis of epilepsy, major depressive disorder, bipolar disorder, schizophrenia or a related disorder, personality disorder, Tourette's disorder, or psychosis not otherwise specified.
3. Currently meeting DSM-5 criteria for autism spectrum disorder, pervasive developmental disorder, obsessive-compulsive disorder, post-traumatic stress disorder, or any other anxiety disorder as the primary diagnosis.
4. Use of anticonvulsants including carbamazepine and valproic acid, antidepressants, mood stabilizers including lithium, benzodiazepines, cholinesterase inhibitors, or any drug known to inhibit CYP2D6 activity within two weeks of Visit 2.
5. Use of herbal supplements within one week of Visit 2.
6. Known or suspected intelligence quotient (IQ) < 70.
7. Unstable endocrinological or neurological conditions which confound the diagnosis or are a contraindication to treatment with antipsychotics.
8. Suicidality, defined as either active suicidal plan/intent or active suicidal thoughts in the six months before the Screening Visit or more than one-lifetime suicide attempt.
9. Pregnancy or refusal to practice contraception during the study (for female subjects of childbearing potential and sexually active males).
10. Substance or alcohol use during the last three months.
11. Urine drug test at screening that is positive for alcohol or drugs of abuse.
12. Known allergy or sensitivity to molindone hydrochloride.
13. Any reason which, in the opinion of the Investigator or the Sponsor, would prevent the subject and subject's caregiver from participating in the study or complying with the study procedures.
14. Use of an investigational drug or participation in an investigational study within 30 days prior to Visit 2.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 333 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azmi Nasser, PhD, Study Director — Supernus Pharmaceuticals, Inc.
Locations (28):
- United States (28):
  - Woodland Research Northwest, Rogers, Arkansas
  - ProScience, Culver City, California
  - Behavioral Research Specialists, Glendale, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - Meridien Research at Florida Clinical Research Center, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Florida Clinical Research Center, LLC., Maitland, Florida
  - CNS Healthcare of Orlando, Orlando, Florida
  - American Medical Research, Chicago, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Hugo W Moser Research Institute at Kennedy Krieger, Baltimore, Maryland
  - Finger Lakes Clinical Research, Rochester, New York
  - Ohio State University Nisonger Center Clinical Trials Program, Columbus, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - CNS Healthcare, Memphis, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Relaro Medical Trials, Dallas, Texas
  - Bayou City Research Corporation, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Road Runner Research, San Antonio, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Aspen Clinical Research, Orem, Utah
  - Alliance Research Group, LLC., Richmond, Virginia
  - Seattle Children's Research Institute, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects were treated with a Placebo
  Placebo
- Low Dose SPN-810 (18 mg): Subjects were treated with a low dose SPN-810 (18 mg)
- High Dose SPN-810 (36 mg): Subjects were treated with a high dose SPN-810 (36 mg)
Period: Overall Study
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
Started (The number of subjects is based on the randomized population that included all those enrolled subjects who complete the Baseline Period, meet the inclusion/exclusion criteria and are randomized.) | 130 | 65 | 138
Intent-to-Treat (The number of subjects is based on the intent-to-treat population (ITT) which include all subjects who received at least 1 dose of study drug and have a baseline and at least 1 valid post-randomization assessment of frequency of IA behaviors based on IA diary entry.) | 125 | 65 | 135
Safety (The number of subjects is based on the Safety Population which includes all randomized subjects who received at least 1 dose of study drug and have at least one post-randomization safety measurements.) | 126 | 65 | 137
Completed (Randomized Population only) | 114 | 58 | 101
Not Completed | 16 | 7 | 37
Not completed — Withdrawal by Subject | 1 | 0 | 4
Not completed — Withdrawal By Parent/Guardian | 5 | 3 | 9
Not completed — Lost to Follow-up | 4 | 2 | 6
Not completed — Adverse Event | 4 | 0 | 10
Not completed — Physician Decision | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Other, Multiple Categories | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: The ITT population includes subjects who received at least 1 dose of study drug and have a baseline and at least 1 valid post-randomization assessment of the frequency of IA behaviors based on IA diary entry.
Groups:
- Placebo: Subjects treated with a Placebo
- Low Dose SPN-810 (18 mg): Subjects treated with low dose of SPN-810
- High Dose SPN-810 (36 mg): Subjects treated with high dose of SPN-810
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg) | Total
Number analyzed (Participants) | 125 | 65 | 135 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (1.95) | 9.1 (1.65) | 9.1 (1.84) | 9.0 (1.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 14 | 34 | 81
  Male | 92 | 51 | 101 | 244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 7 | 19 | 46
  Not Hispanic or Latino | 104 | 57 | 116 | 277
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 4 | 7
  Asian | 0 | 0 | 1 | 1
  Black or African American | 21 | 26 | 39 | 86
  White | 94 | 35 | 85 | 214
  Other | 8 | 3 | 6 | 17
Retrospective-Modified Overt Aggression Scale (R-MOAS) [Mean (Standard Deviation); unit: units on a scale] — R-MOAS scale gauges the severity of aggressive behavior: the frequency of the 16 behaviors is rated over the past week in 4 areas (a-d). For each open question in each area, the parent rates the aggressive behaviors on a scale from 0 to 5 or more times. To each area corresponds a weighted category: 1(a), 4(b), 2(c) and 3(d). Therefore, the sum of each area yields a maximum weighted score of 20 (a), 120 (b), 60 (c) and 90 (c). The total score is the sum of the four area scores or 0-290, the higher the score, the more severe the aggressive behavior is.
  units on a scale | 69.70 (33.277) | 73.82 (37.552) | 66.64 (30.966) | 69.25 (33.257)
Vitiello Aggression Scale [Mean (Standard Deviation); unit: units on a scale] — The Vitiello Aggression Scale is a 10-item rating scale that uses a cluster analysis to categorize aggression into two subtypes; predatory and affective. The predatory score is calculated by summing up the individual scores from items 2, 5, 7, 9, and 10. The affective score is calculated by summing up the individual scores from items 1, 3, 4, 6, and 8.The total score is the difference of predatory score and affective score. Possible range of total score varies from 5 (completely predatory) to -5 (completely affective).
  units on a scale | -3.65 (1.042) | -3.57 (1.145) | -3.42 (1.018) | -3.54 (1.055)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy and Safety of SPN-810 on the Frequency of Impulsive Aggression (IA) Measured by the Impulsive Aggression Diary
Description: The primary efficacy endpoint was percent change (PCHT) in the frequency (unweighted score) of IA behaviors per 7 days in the treatment (titration and maintenance) period relative to the Baseline period calculated over the number of days with non-missing IA diary data. PCHT was then calculated as 100 x (T - B)/B, where T and B are IA behavior frequencies per 7 days during the treatment period (from Day 2 through Visit 6, inclusive) and baseline period (Day ≤1), respectively. The IA behavior frequency per 7 days is defined as (SUM/DAY) x 7, where SUM is the total of the IA behaviors reported in the subject IA diary, and DAY is the number of days with a non-missing IA score in the subject IA diary during the specified study period.
Time Frame: Daily measure from Visit 2 (Week-2) to Visit 6 (Week 5) for a total of 7 weeks
Population: Intent-to-Treat (ITT) Population: The ITT population includes subjects who received at least 1 dose of the study drug and have a baseline and at least 1 valid post-randomization assessment of the frequency of IA behaviors based on IA diary entry.
Measure: Median (Full Range); unit: percent change of IA behaviors
Groups:
- Low Dose SPN-810 (18 mg): Subjects treated with a low dose of SPN-810
- High Dose SPN-810 (36 mg): Subjects treated with a high dose of SPN-810
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 125 | 65 | 135
percent change of IA behaviors | -48.16 [-100.0 to 98.3] | -47.88 [-97.4 to 57.3] | -58.56 [-100.0 to 140.5]
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); Test type: Superiority; p = 0.0916, Wilcoxon (Mann-Whitney); Median Difference (Net) = -7.08, 95% CI 2-sided [-15.38 to 1.22]
Statistical Analysis 2: Comparison: Placebo vs Low Dose SPN-810 (18 mg); Based on the results of a prespecified interim analysis, the enrollment of the low dose SPN-810 arm was halted, and this treatment arm was dropped. Accordingly, all analysis of primary and secondary endpoints focused on the comparison of SPN-810 high dose and placebo; Test type: Superiority; p = 0.7136, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.76, 95% CI 2-sided [-11.78 to 8.27]

2. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by Clinical Global Impression-Improvement (CGI-I) Scale Investigator Rated
Description: The Clinical Global Impression - Improvement Scale (CGI-I) is an assessment of how much the patient's illness has improved or worsened relative to a baseline state at the beginning of treatment.
  CGI-I was evaluated by the Investigator at each visit on a 7-point scale with 1=very much improved, 2= much improved, 3= minimally improved, 4= no change, 5= minimally worse, 6= much worse, 7= very much worse
Time Frame: Visit 4 (Week 1), Visit 5 (Week 2) and Visit 6 (Week 5), a total of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Subjects treated with Placebo
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 125 | 65 | 135
score on a scale
  Visit 4: number analyzed (Participants) | 121 | 65 | 134
  Visit 4 | 3.28 (0.829) | 3.14 (0.933) | 3.03 (0.867)
  Visit 5: number analyzed (Participants) | 118 | 64 | 120
  Visit 5 | 2.92 (0.935) | 2.81 (1.006) | 2.68 (0.970)
  Visit 6: number analyzed (Participants) | 112 | 57 | 101
  Visit 6 | 2.72 (0.979) | 2.58 (1.101) | 2.43 (0.983)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); Test type: Superiority — This analysis pertains to Visit 4; p = 0.0238, Mixed Models Analysis; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.46 to -0.03], Standard Error of Mean 0.108
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 5; Test type: Superiority; p = 0.0683, Mixed Models Analysis; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.47 to 0.02], Standard Error of Mean 0.123
Statistical Analysis 3: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 6; Test type: Superiority; p = 0.0742, Mixed Models Analysis; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.51 to 0.02], Standard Error of Mean 0.136

3. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by Clinical Global Impression - Severity Scale (CGI-S)
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a single item clinician rating of clinician's assessment of the severity of IA behaviors CGI-S was evaluated by the Investigator at each visit on a 7- point scale with 1=Normal, 2=Borderline ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Extremely ill Data represent the change between Baseline (Visit 3/Day 1) and three time points: Visit 4 (Week 1); Visit 5 (Week 2) and Visit 6 (Week 5).
Time Frame: Baseline/Visit 3 (Day 1), Visit 4 (Week 1), Visit 5 (Week 2), and Visit 6 (Week 5). The total duration of the study was 5 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 125 | 65 | 135
score on a scale
  Visit 4: number analyzed (Participants) | 122 | 65 | 134
  Visit 4 | -0.55 (0.772) | -0.71 (0.964) | -0.65 (0.928)
  Visit 5: number analyzed (Participants) | 118 | 64 | 120
  Visit 5 | -0.88 (0.953) | -1.08 (1.238) | -1.08 (1.081)
  Visit 6: number analyzed (Participants) | 113 | 58 | 102
  Visit 6 | -1.13 (1.106) | -1.29 (1.325) | -1.37 (1.080)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); Test type: Superiority — This analysis pertains to Visit 4; p = 0.3713, Mixed Models Analysis; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.30 to 0.11], Standard Error of Mean 0.105
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 5; Test type: Superiority; p = 0.1367, Mixed Models Analysis; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.45 to 0.06], Standard Error of Mean 0.131
Statistical Analysis 3: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 6; Test type: Superiority; p = 0.1729, Mixed Models Analysis; Median Difference (Net) = -0.20, 95% CI 2-sided [-0.49 to 0.09], Standard Error of Mean 0.146

4. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by Child Health Questionnaire Parent Form 28-item (CHQ-PF28)
Description: CHQ-PF28) is a short generic measure of health status and health-related quality of life. The 28 items have 4, 5, or 6 response options, divided over 8 multi-item scales (physical functioning, general behavior, mental health, self-esteem, general health perceptions, parental impact: emotional, parental impact: time, and family activities) and 5 single item concepts (role functioning: emotional/behavior, role functioning: physical, bodily pain, family cohesion, and change in health). In addition, the individual scale scores will be aggregated to derive 2 summary component scores: the physical functioning and psychosocial health summary scores. The range on subscales and the overall scale is 0-100 (0 = worst possible health state; 100 = best possible health state). Data represent the change from Baseline (Visit 3) one time point, Visit 6 (Week 5).
Time Frame: Baseline Visit 3 (Day 1) and Visit 6 (Week 5). Total duration of the study was 5 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Subjects treated with a Placebo
  Placebo
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 125 | 65 | 135
score on a scale
  Physical Functioning Summary Score At Visit 6: number analyzed (Participants) | 113 | 58 | 101
  Physical Functioning Summary Score At Visit 6 | 8.52 (10.786) | 10.11 (11.351) | 9.53 (11.199)
  Psychosocial Health Summary Score At Visit 6: number analyzed (Participants) | 113 | 58 | 101
  Psychosocial Health Summary Score At Visit 6 | -0.99 (7.466) | -2.66 (7.200) | -2.09 (7.587)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the physical functioning summary score at Visit 6; Test type: Superiority; p = 0.1407, ANCOVA; Mean Difference (Net) = 2.15, 95% CI 2-sided [-0.72 to 5.02], Standard Error of Mean 1.456
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the psychosocial health summary score at Visit 6; Test type: Superiority; p = 0.5586, ANCOVA; Mean Difference (Net) = -0.53, 95% CI 2-sided [-2.29 to 1.24], Standard Error of Mean 0.898

5. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by Parenting Stress Index, Fourth Edition, Short Form (PSI-4-SF)
Description: The PSI-4-SF is a 36-item self-report measure of parenting stress. Three subscales Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC) consist of 12 items each. Parent chooses one of the 5 responses against each item. The 5 responses are: Strongly Agree (SA), Agree (A), Not Sure (NS), Disagree (D), and Strongly Disagree (SD) to indicate the degree to which they agree with each statement. The PD subscale raw score ranges from 12-60, P-CDI and DC each subscale raw score ranges from 16-56. The total stress raw score is the sum of the three subscales (PD+P-CDI+ DC) with a minimum score of 44 and a maximum score of 172. The total stress score is then converted into the percentile score. Parents with a 91st percentile or higher are experiencing clinically significant levels of stress. Data represent the change between Baseline (Visit 3) and one time point, Visit 6 (Week 5).
Time Frame: Baseline Visit 3 (Day 1) and Visit 6 (Week 5). Total duration of the study was 5 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- High Dose SPN-810 (36 mg): Subjects treated with a high dose of SPN-810
  SPN-810
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 125 | 65 | 135
score on a scale
  Total Score at Visit 6: number analyzed (Participants) | 111 | 58 | 102
  Total Score at Visit 6 | -8.95 (15.539) | -5.52 (15.030) | -8.40 (16.015)
  Parental Distress Domain at Visit 6: number analyzed (Participants) | 112 | 58 | 102
  Parental Distress Domain at Visit 6 | -1.96 (7.049) | -1.95 (6.163) | -2.00 (7.319)
  Parent-Child Dysfunctional Interaction Domain at Visit 6: number analyzed (Participants) | 111 | 58 | 102
  Parent-Child Dysfunctional Interaction Domain at Visit 6 | -2.94 (6.413) | -1.43 (6.623) | -2.69 (6.617)
  Difficult Child Domain at Visit 6: number analyzed (Participants) | 112 | 58 | 102
  Difficult Child Domain at Visit 6 | -4.21 (7.193) | -2.14 (5.766) | -3.72 (5.598)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Total Stress summary score Visit 6; Test type: Superiority; p = 0.7637, ANCOVA; Median Difference (Net) = -0.62, 95% CI 2-sided [-4.70 to 3.45], Standard Error of Mean 2.070
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Parental Distress Domain score at Visit 6; Test type: Superiority; p = 0.8365, ANCOVA; Mean Difference (Net) = -0.18, 95% CI 2-sided [-1.95 to 1.58], Standard Error of Mean 0.895
Statistical Analysis 3: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Parent-Child Dysfunctional Interaction score at Visit 6; Test type: Superiority; p = 0.4606, ANCOVA; Mean Difference (Net) = -0.61, 95% CI 2-sided [-2.24 to 1.02], Standard Error of Mean 0.829
Statistical Analysis 4: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Difficult Child Domain score Visit 6; Test type: Superiority; p = 0.8222, ANCOVA; Mean Difference (Net) = -0.19, 95% CI 2-sided [-1.84 to 1.46], Standard Error of Mean 0.837

6. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by the Caregiver Clinical Global Impression - Improvement Scale (CGI-I)
Description: The CGI scale was developed to provide a brief, stand-alone assessment of the clinician's view of a subject's global functioning prior to and after administration of a study medication. The scale was also rated by the caregiver to assess the improvement of IA behaviors.
  CGI-I was evaluated by the Caregiver at each visit on a 7-point scale with 1=very much improved, 2= much improved, 3= minimally improved, 4= no change, 5= minimally worse, 6= much worse, 7= very much worse
Time Frame: Visit 4 (Week 1), Visit 5 (Week 2) and Visit 6 (Week 5), a total of 4 weeks]
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 125 | 65 | 135
score on a scale
  Visit 4: number analyzed (Participants) | 122 | 65 | 133
  Visit 4 | 3.11 (0.986) | 3.12 (1.008) | 2.91 (0.917)
  Visit 5: number analyzed (Participants) | 118 | 63 | 120
  Visit 5 | 2.93 (0.967) | 2.76 (1.043) | 2.61 (1.087)
  Visit 6: number analyzed (Participants) | 112 | 58 | 101
  Visit 6 | 2.66 (1.205) | 2.64 (1.210) | 2.29 (1.117)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); Test type: Superiority — This analysis pertains to Visit 4; p = 0.1031, Mixed Models Analysis; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.43 to 0.04], Standard Error of Mean 0.121
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); Test type: Superiority — This analysis pertains to Visit 5; p = 0.0250, Mixed Models Analysis; Mean Difference (Net) = -0.30, 95% CI 2-sided [-0.56 to -0.04], Standard Error of Mean 0.132
Statistical Analysis 3: Comparison: Placebo vs High Dose SPN-810 (36 mg); Test type: Superiority — This analysis pertains to Visit 6; p = 0.0384, Mixed Models Analysis; Mean Difference (Net) = -0.33, 95% CI 2-sided [-0.64 to -0.02], Standard Error of Mean 0.158

7. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by the Swanson, Nolan, Pelham Rating Scale- Revised (SNAP-IV) Rating Scale
Description: The Swanson, Nolan, Pelham Rating Scale-Revised (SNAP-IV) includes 18 ADHD and 8 oppositional defiant disorder (ODD) symptoms. The symptoms are scored on a 4-point scale. The ratings from the SNAP-IV scale are grouped into the following 4 subscales: ADHD Inattention (items #1-9), ADHD Hyperactivity/Impulsivity (items#10-18), ODD (items# 19-26), and ADHD-combined (first two scales combined, items #1-18). Each subscale score is the average rating of the items scores for the subscale. Therefore, for the inattention, the hyperactivity/impulsivity and the combined subscales the scores range from 0-27, while for the ODD scores range from 0-24; the higher is the score, worsen is the outcome. The following average cut-off are considered clinically significant based on the 95th percentile: 1.78 (Inattention items), 1.44 (hyperactivity/impulsivity items), 1.88 (ODD items) and 1.67 (combined type). Data represent the change between Baseline (Visit 3) and the end of the study, Visit 6 (Week 5).
Time Frame: Baseline Visit 3 (Day 1) and Visit 6 (Week 5). Total duration of the study was 5 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 125 | 65 | 135
score on a scale
  Inattention subscale: number analyzed (Participants) | 113 | 58 | 102
  Inattention subscale | -0.45 (0.606) | -0.50 (0.742) | -0.53 (0.661)
  Hyperactivity/Impulsivity subscale: number analyzed (Participants) | 113 | 58 | 102
  Hyperactivity/Impulsivity subscale | -0.43 (0.661) | -0.50 (0.721) | -0.59 (0.756)
  Oppositional Defiant Disorder subscale: number analyzed (Participants) | 113 | 58 | 102
  Oppositional Defiant Disorder subscale | -0.50 (0.698) | -0.54 (0.833) | -0.58 (0.838)
  Combined subscale: number analyzed (Participants) | 113 | 58 | 102
  Combined subscale | -0.44 (0.576) | -0.50 (0.677) | -0.56 (0.657)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the inattention subscale at Visit 6; Test type: Superiority; p = 0.1935, ANCOVA; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.27 to 0.06], Standard Error of Mean 0.084
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to hyperactivity/Impulsivity subscale at Visit 6; Test type: Superiority; p = 0.1445, ANCOVA; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.32 to 0.05], Standard Error of Mean 0.092
Statistical Analysis 3: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the oppositional defiant disorder subscale at Visit 6; Test type: Superiority; p = 0.1064, ANCOVA; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.36 to 0.03], Standard Error of Mean 0.100
Statistical Analysis 4: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the combined scale score at Visit 6; Test type: Superiority; p = 0.1418, ANCOVA; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.28 to 0.04], Standard Error of Mean 0.082

ADVERSE EVENTS:
Time Frame: Visit 3 (Day 1) to Visit 7 (Week 6)-End of Study, a total of 6 weeks
Description: Adverse events reporting pertains to the Safety Population which include all randomized subjects who received at least 1 dose of study drug and have at least one post-randomization safety measurements.
Groups:
- Placebo: Subjects were treated with a Placebo
- Low Dose SPN-810 (18 mg): Subjects were treated with a low dose of SPN-810
- High Dose SPN-810 (36 mg): Subjects were treated with a high dose of SPN-810
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/65 | 0/137
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/65 | 2/137
Other Adverse Events (participants affected / at risk) | 18/126 | 10/65 | 26/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=126) | Low Dose SPN-810 (18 mg) (N=65) | High Dose SPN-810 (36 mg) (N=137)
Vision blurred (Eye disorders) | 0 | 0 | 1
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=126) | Low Dose SPN-810 (18 mg) (N=65) | High Dose SPN-810 (36 mg) (N=137)
Fatigue (General disorders) | 1 | 2 | 10
Headache (General disorders) | 2 | 2 | 7
Increased appetite (Metabolism and nutrition disorders) | 6 | 0 | 9
Blood prolactin Increased (Investigations) | 1 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 2 | 2

LIMITATIONS AND CAVEATS:
There were no limitations or caveats with the clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT02618408/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT02618408/SAP_001.pdf